CLINICAL TRIAL: NCT00006380
Title: Phase I Evaluation of 131I-J591 Murine Monoclonal Antibody in Patients With Progressive Androgen-Independent Prostate Cancer
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-061; CDR0000068254 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1870
Record Dates: First submitted 2000-10-04; First posted 2004-06-09 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Biological: monoclonal antibody muJ591
Radiation: iodine I 131 monoclonal antibody muJ591

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have prostate cancer that no longer responds to antiandrogen therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the biodistribution and normal organ dosimetry of iodine I 131 monoclonal antibody muJ591 in patients with progressive androgen independent prostate cancer. II. Determine the safety of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients. IV. Determine the human antimouse antibody response in these patients to this drug. V. Determine the antitumor effects of this drug in these patients.

OUTLINE: This is a dose escalation study of iodine I 131 monoclonal antibody muJ591 (131I-J591). Patients receive unlabeled monoclonal antibody muJ591 IV over 1 hour followed by 131I-J591 IV over 1 hour. Cohorts of 3-6 patients receive escalating doses of 131I-J591 (radioactivity is escalated, monoclonal antibody dose is fixed) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 6 patients experience dose limiting toxicity. Patients are followed at weeks 3, 4, 6, 8, 9, and 12, and then every 6 months until month 21.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed androgen independent prostate cancer that is progressing under castrate levels of testosterone Progression documented in one of the following ways: A minimum of 3 rising PSA values from baseline obtained 1 week or more apart or 2 measurements 2 weeks or more apart New osseous lesions on bone scan Greater than 25% increase in bidimensionally measurable soft tissue disease, or the appearance of new sites of disease Patients on an antiandrogen must have shown progression off of the antiandrogen prior to study Testosterone no greater than 50 ng/mL No residual proctitis following radiotherapy No active CNS or epidural primary tumor or metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC greater than 3,500/mm3 Hemoglobin greater than 10 g/dL Platelet count greater than 150,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL GGT less than upper limit of normal (ULN) AST less than ULN PT less than 14 seconds No autoimmune hepatitis Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No New York Heart Association class III or IV cardiac disease Pulmonary: No severe debilitating pulmonary disease Other: No active uncontrolled infection or infection requiring IV antibiotic treatment No evidence of human antimouse antibody No prior autoimmune disease No prior GI hemorrhage HIV negative Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 months since prior packed red blood cell transfusion No prior murine or human antibody therapy No prior murine protein No other concurrent immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy and recovered No concurrent chemotherapy Endocrine therapy: See Disease Characteristics Concurrent gonadotropin releasing hormone analogs required for patients who have not undergone surgical orchiectomy No other concurrent hormonal therapy Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy and recovered No prior diagnostic scintigram (e.g., ProstaScint, Myoscint, or Oncoscint) No prior radiotherapy to more than the sternum alone OR No primary radiotherapy to the prostate and one other site OR No prior radiotherapy to more than 25% of the skeleton No prior treatment with strontium chloride Sr 89 or Samarium Sm 153 lexidronam pentasodium No concurrent radiotherapy to localized sites (e.g.,bone) used as indicator lesions Surgery: No concurrent surgery to sole site of measurable disease Other: At least 4 weeks since investigational anticancer therapeutic drugs and recovered No concurrent aspirin, nonsteroidal antiinflammitory agents, anticoagulants, or other drugs that may induce or exacerbate a bleeding tendency

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard I. Scher, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States